CLINICAL TRIAL: NCT03934034
Title: A Prospective Registry For Patients With Non-Tuberculous Mycobacterial (NTM) Pulmonary Disease in Korea.
Acronym: NTM-KOREA
Status: Not yet recruiting | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Collaborators: Asan Medical Center (Other); Samsung Medical Center (Other); Pusan National University Hospital (Other); Severance Hospital (Other); Pusan National University Yangsan Hospital (Other); Chonnam National University Hospital (Other); Korean Institute of Tuberculosis (Other); International Tuberculosis Research Center (Other)
Responsible Party: Principal Investigator, Jae-Joon Yim, Professor, Pulmonary and Critical Care Medicine, Seoul National University Hospital
Other Study IDs: NTM-KOREA
Record Dates: First submitted 2019-04-22; First posted 2019-05-01 (Actual); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: Pulmonary Disease; Pulmonary Infection; Non-Tuberculous Mycobacterial Pneumonia
Keywords: NTM; Registry; Pulmonary infection
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The incidence and prevalence of pulmonary disease due to Non-tuberculous mycobacteria (NTM) is increasing worldwide, and this trend has been confirmed in Korea. Treatment of NTM pulmonary disease is difficult and usually requires more than two years of long-term treatment, and the antibiotic regimens used in treatment vary. Therefore, it is difficult to track the natural history of patients with NTM pulmonary disease, to evaluate the treatment outcome, and to understand the effect of specific medicines on the outcome. Establishing a prospective registry of patients with NTM pulmonary disease is expected to accurately evaluate the progress, treatment modality, and treatment outcome of NTM pulmonary disease.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of NTM pulmonary disease.
2. The causative agent of NTM pulmonary disease includes: M. avium complex, or M. abscessus subspecies abscessus, or M. abscessus subspecies massiliense, or M. kansasii.
3. Patients who starts new treatment (those who have previous history of treatment are eligible)

Exclusion Criteria

1. Patients who have been treated for more than 4 weeks.
2. The causative agent of NTM pulmonary disease is none of M. avium complex, M. abscessus subspecies abscessus, M. abscessus subspecies massiliense, or M. kansasii.

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with NTM lung disease initiating treatment at each hospital participating in the study
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-04 (Estimated); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Treatment success rate | Through study completion, at 1 year after treatment start at enrollment
  Analysis of treatment success rate according to species of NTM lung disease patients in Korea

SECONDARY OUTCOMES:
Comparison of the efficacy among different regimens for the treatment of certain species of NTM | Through study completion, at 1 year after treatment start at enrollment
  Comparison of the outcomes measured by culture conversion among different regimens for the treatment of certain species of NTM
Number of participants with changing culture results during treatment | Through study completion, at 1 year after treatment start at enrollment
  Number of participants with changing culture results during treatment
Number of participants with treatment-related adverse events | Through study completion, at 1 year after treatment start at enrollment
  Number of participants with treatment-related adverse events specifically described in the protocol

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kwak N, Henkle E, Hwang H, Jeon D, Jhun BW, Jo KW, Kang YA, Kim HJ, Kim JY, Kim YR, Kwon YS, Lee JH, Mok J, Park Y, Shim TS, Sohn H, Whang J, Yim JJ. Improvement in Health-Related Quality of Life Following Antibiotic Treatment in Nontuberculous Mycobacterial Pulmonary Disease: Initial Analysis of the NTM-KOREA Cohort. Clin Infect Dis. 2024 Jun 14;78(6):1690-1697. doi: 10.1093/cid/ciae131. PMID 38563246